CLINICAL TRIAL: NCT00942513
Title: Effect of Lactose, Fructose, Sucrose, Whey Protein, and Soy Protein on Substrate Absorption and Oxidation: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: David J. Baer, Ph. D., Principal Investigator, USDA_ARS
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 2007-342
Record Dates: First submitted 2009-07-17; First posted 2009-07-21 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Substrate Absorption; Substrate Oxidation; Glucose Regulation
Keywords: substrate absorption; substrate oxidation; glucose regulation; whey protein; soy protein; sucrose; fructose; lactose
MeSH Terms: interventions — 2-(9H-fluoren-9-yl)methoxycarbonylamino-3-ethoxy-N-tritylsuccinamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: trt 1 — Fructose - 14 g; Lactose - 10 g; Sucrose - 16 g; Starch - 40 g; Whey Protein Isolate - 40 g; Soy Protein Isolate - 0 g
Other: trt 2 — Fructose - 30 g; Lactose - 10 g; Sucrose - 0 g; Starch - 40 g; Whey Protein Isolate - 40 g; Soy Protein Isolate - 0 g
Other: trt 3 — Fructose - 24 g; Lactose - 8 g; Sucrose - 8 g; Starch - 40 g; Whey Protein Isolate - 40 g; Soy Protein Isolate - 0 g
Other: trt 4 — Fructose - 0 g; Lactose - 0 g; Sucrose - 40 g; Starch - 40 g; Whey Protein Isolate - 40 g; Soy Protein Isolate - 0 g
Other: trt 5 — Fructose - 0 g; Lactose - 0 g; Sucrose - 40 g; Starch - 40 g; Whey Protein Isolate - 0 g; Soy Protein Isolate -40 g
Other: trt 6 — Fructose - 0 g; Lactose - 40 g; Sucrose - 0 g; Starch - 40 g; Whey Protein Isolate - 40 g; Soy Protein Isolate - 0 g
Other: trt 7 — Fructose - 0 g; Lactose - 40 g; Sucrose - 0 g; Starch - 40 g; Whey Protein Isolate - 0 g; Soy Protein Isolate -40 g

SUMMARY:
Does the consumption of various combinations of mono and disaccharides (lactose, sucrose and fructose) and protein isolates (whey or soy) result in altered substrate absorption, substrate oxidation, and glucose regulation? This proposed research will provide data to determine the relative contribution of source of protein (whey vs soy) and carbohydrate (mono- and disaccharides) on the observed effects of dairy products on absorption, substrate oxidation and glucoregulation mechanisms that affect body composition.

DETAILED DESCRIPTION:
Epidemiological research has shown that dairy products aid in weight loss and weight maintenance. Some evidence suggests that this effect is due to the whey component (which contains whey proteins and lactose) of milk. Previous work from our laboratory has demonstrated that chronic administration of whey protein concentrate results in decreased body fat and insulin concentration. Recent research (unpublished) from Castonguay and colleagues (University of Maryland, College Park, MD) has suggested that specific combinations of sucrose, maltose and lactose similarly alter body fat levels in rats. This proposed research will provide data to determine the relative contribution of source of protein (whey vs soy) and carbohydrate (mono- and disaccharides) on the observed effects of dairy products on absorption, substrate oxidation and glucoregulation mechanisms that affect body composition.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* BMI at least 20 and less than 38 kg/m2 and body weight < 300 lbs.
* Age 25 to 65 years at beginning of study.
* Fasting glucose < 126 mg/dL.
* Blood pressure < 160/100 mm Hg.
* Total plasma cholesterol < 280 mg/dL.
* Nonsmokers or tobacco users (for at least 6 months prior to the start of the study.)

Exclusion Criteria:

* History or presence of kidney disease, liver disease, gout, certain cancers, thyroid disease, gastrointestinal, other metabolic diseases, or malabsorption syndromes.
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin.
* History of eating disorders.
* Volunteers who routinely participate in heavy exercise or volunteers who initiate an exercise program during the study.
* Volunteers who have lost 10% of body weight within the last 12 months .
* Volunteers who have been on Atkins, South Beach or similar diet in 3 months prior to start of study.
* Use of prescription or over-the-counter antiobesity medications or supplements (e.g., phenylpropanalamine, ephedrine, caffeine, during and for at least 6 months prior to the start of the study).
* Known (self-reported) allergy or adverse reaction to dairy products (including lactose) or soy.
* Volunteers who consume whey or soy protein supplements.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Baer, Ph. D., Principal Investigator — United States Department of Agriculture (USDA)
Locations (1):
- USDA-ARS, Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States